CLINICAL TRIAL: NCT00703235
Title: Intravitreal Bevacizumab for Diabetic Macular Edema
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Isfahan Ophthalmology Research Center (Network)
Other Study IDs: MUI - clinical - 185290
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2008-06-23 (Estimated); Status verified 2008-06

CONDITIONS: Macular Edema; Diabetic Retinopathy
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab

SUMMARY:
Diabetic macular edema is a common cause of visual loss among diabetic patients. Studies have demonstrated the role of vascular endothelial growth factor (VEGF) in the pathogenesis of edema.

This study designed to evaluate the effect of Intravitreal injection of a recombinant monoclonal anti-VEGF antibody, Bevacizumab, for treatment of diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Clinically significant macular edema
* Possibility of performing macular OCT
* Consent of patient for inclusion in the study

Exclusion Criteria:

* History of macular photocoagulation in less than 6 months of inclusion in the study
* Necessity of surgical intervention
* Rejection of the remaining in the study by patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult